CLINICAL TRIAL: NCT02111070
Title: Open-label, Phase I Clinical Trial to Assess the Immunogenicity and Safety of the 'IL-YANG Inactivated Split Influenza Vaccine' in Healthy Korean Male Subjects
Brief Title: Immunogenicity and Safety Study of Inactivated Split Influenza Vaccine' in Healthy Korean Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IY_IFEZ_101
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Influenza; Influenza vaccine; Split influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ILYANG Inactivated split influenza vaccine (Experimental): IL-YANG FLU Vaccine Vial INJ 0.5mL by intramuscular injection
  Interventions: Biological: IL-YANG FLU Vaccine

INTERVENTIONS:
Biological: IL-YANG FLU Vaccine — 0.5mL

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of IL-YANG Inactivated Split Influenza Vaccine (IL-YANG FLU Vaccine Vial INJ.) administered as a single intramuscular injection

DETAILED DESCRIPTION:
This was an open-label study. Subjects providing voluntary written informed consent underwent protocol-specific assessments and tests within 4 weeks prior to administration of the study vaccine, and those who met all of the inclusion/exclusion criteria and were considered eligible were sequentially enrolled in the study.

Subjects enrolled in the study received 0.5ml of the study vaccine as an intramuscular injection in the deltoid muscle, and returned to the clinic every day for the first 3 days. On Day 14 post-vaccination, subjects underwent the safety assessments. On Day 28 post-vaccination, subjects returned for safety and immunogenicity assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between 20 and 55 years of age at screening
* Body weight of ≥ 55kg and within ±20% of ideal body weight (ideal body weight = (height cm - 100) X 0.9) at screening
* Subjects with no congenital or chronic disease who were considered suitable for the study after screening assessments (investigator's opinion, medical history, physical examination, laboratory test, chest X-ray, and ECG) conducted within 28 days prior to vaccination
* Subjects who were given, and fully understood, the information about the study, made a voluntary decision, and provided written informed consent, to participate in the study and comply with all applicable study requirements

Exclusion Criteria:

* Subjects with pre-vaccination HI antibody titer ≥ 1:40
* Subjects who have known or suspected infection with HAV, HBV, HCV, HIV or VDRL (via ELISA screening or medical history taking)
* Subjects who have concurrent or a past history of immune deficiency disease
* Subject who had participated in blood donation within 1 week prior to vaccination, or are planning to participate in blood donation from Day 1 until Month 7 post-vaccination
* Subject with a history of Guillain-Barre syndrome
* Subject with hemophilia, thrombocytopenia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subjects who have concurrent or a past history of, malignant tumor of internal organ or blood vessels or skin metastasis
* Subjects with known allergy to a drug, food or latex, who had a history of anaphylaxis
* Subjects who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine or symptoms of suspected acute disease within 14 days prior to administration of the study vaccine
* Subjects who received another experimental drug or vaccine within 28 days before administration of the study vaccine or are planning to receive another experimental drug or vaccine during the study.
* Subjects who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or are expecting to be treated with immunoglobulin or blood-derived products during the study
* Subjects who had received, or are scheduled to receive, systemic immunosuppressive therapy, radiation therapy or high-dose steroid therapy within the last 6 months prior to administration of the study
* Subjects who had received, or are expected to receive, the medications listed below: Within 28 days prior to administration of the study vaccine: Oriental herbal medicine, Within 14 days prior to administration of the study vaccine: Prescription drugs, Within 7 days prior to administration of the study vaccine: Over-the-counter medicine (including vitamin/mineral supplements)
* Subjects with a history of, or suspected, drug abuse (amphetamine, barbiturates, opioids, benzodiazepines, etc.) based on subject interview and physical examination.
* Subjects with excessive consumption of caffeine (> 5 cups/day) and alcohol (>3 units/day, 1unit= 10g or 12.5ml of pure alcohol), and excessive smoking (>10 cigarettes/day)
* Subject with a known allergy to eggs, chicken, or any components of the study vaccine
* Subjects who in the investigator's opinion, may not be suitable for vaccination or who may interfere with the objective assessment of the study outcomes.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Solicited local & general AE, Unsolicited AE | up to Day28(+7)
  Solicited local reaction: pain, tenderness, redness, swelling Solicited general reactions: fever, nausea/vomiting, diarrhea, headache, fatigue, myalgia
Percentage of subjects achieving seroprotection for HI antibody after administration of the study vaccine | Day28(+7)
  Seroprotection: HI antibody titer ≥ 1:40 28 days after the administration of the study vaccine

SECONDARY OUTCOMES:
GMT of HI antibody titer before vaccination and after vaccination | Day28(+7)
  GMT(Geometric Mean Titer) and GMR(Geometric Mean Ratio), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer
Percentage of subjects with a pre-vaccination (Day 0) HI antibody titer < 1:40, and a minimum four-fold rise in post-vaccination (vaccination + 28 days) HI antibody titer | Day28(+7)
Vital signs measurements, physical examination findings, ECG results, and laboratory measurements (hematology, biochemistry and urinalysis) | Day28(+7)

CONTACTS AND LOCATIONS:
Overall Officials: IL-YANG PHARM, Study Director — IL-YANG Pharmaceutical Co.,LTD
Locations (1):
- Seoul St. Mary's Hospital,The Catholic University of Korea, Seoul, South Korea